CLINICAL TRIAL: NCT04467294
Title: Prospective Register on the Etiologies of Cardiogenic Shock and Their Prognosis at One Year.
Acronym: cardiac shock
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-29; 2019-A01294-53 (Other: IDRCB)
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Cardiogenic Shock
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiogenic shock (CC) is one of the major challenges of current cardiology. Despite the difficulty of establishing a strict and consensual definition, it is accepted that the CC clinically corresponds to persistent hypotension (systolic blood pressure 90 mmHg for at least 30 minutes or need for vasopressor support) associated with signs of visceral hypoperfusion (confusion, mottling, oliguria, hyperlactatemia), and hemodynamic with a lowered heart index ( 1.8 L/min/m2) despite appropriate or high filling pressures. This definition of the European Society of Cardiology (ESC) masks however the great variability of hemodynamic tables grouped under the term of CC and severity levels, also variable.However, it was suggested that the etiology of CC influenced both its hemodynamic profile and therefore its therapeutic management but also its prognosis in the medium and long term.

DETAILED DESCRIPTION:
CC diagnosis remains difficult to carry on admission and is sometimes delayed. Therefore, we would like to compare hemodynamic data from patients with CC status to those admitted for acute heart failure (ICA) to determine if a hemodynamic variable at entry would facilitate the diagnosis of CC.

ELIGIBILITY:
Inclusion Criteria:

* Patients in Cardiac Shock :
* 90 mmHg hypotension or requiring inotropic or vasopressor support,
* owered cardiac output ( 1.8 L/min/m2) to trans-thoracic cardiac ultrasound with high or normal filling pressures
* peripheral hypoperfusion. patients admitted for acute heart failure (ICA) (Acute pulmonary edema chart or left congestive heart failure without CC sign and with ultrasound FEVG at entry 40%.)

Exclusion Criteria:

* Pregnant or nursing women
* Age 18 years
* Person of full age under guardianship
* Staying in a health or social facility
* Person not covered by a social security scheme
* Person deprived of liberty
* Shocks from other etiologies
* Patient with initial cardiac arrest
* Patient with cardiogenic shock due to right ventricular dysfunction
* Patient with pulmonary embolism
* Patient with tamponade
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in Cardiac Shock and patients admitted for acute heart failure (ICA)
Sampling Method: Non-Probability Sample
Enrollment: 1650 (Estimated)
Dates: Start 2020-04-04 (Actual); Primary Completion 2023-04-04 (Estimated); Study Completion 2023-10-04 (Estimated)

PRIMARY OUTCOMES:
prevalence of Cardiac Shock | 12 months

SECONDARY OUTCOMES:
mortality | one month
mortality | one year

CONTACTS AND LOCATIONS:
Overall Officials: Garrido-pradalie Emilie, Study Director — ASSISTANCE PUBLIQUE HÔPITAUX DE MARSEILLE
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, PACA, France

IPD SHARING:
Plan to Share IPD: No